CLINICAL TRIAL: NCT04445519
Title: Phase 3, Randomized, Adaptive Dose-Selection, Multi-regional, Double-Masked, Parallel-Group, 3-Month Trial Evaluating the Safety and Efficacy of NCX 470 vs. Latanoprost 0.005% in Subjects With Open-Angle Glaucoma or Ocular Hypertension (Mont Blanc)
Brief Title: Phase 3 Trial of NCX 470 vs. Latanoprost in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Acronym: Mont Blanc
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nicox Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCX-470-02
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-03

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-masked
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- NCX 470 0.065% (Experimental): NCX 470 Ophthalmic Solution, 0.065% dosed once daily to both eyes (initial phase of trial)
  Interventions: Drug: NCX 470 0.065% (initial phase of trial)
- NCX 470 0.1% (Experimental): NCX 470 Ophthalmic Solution, 0.1% dosed once daily to both eyes (initial phase of trial)
  Interventions: Drug: NCX 470 0.1% (initial phase of trial)
- Latanoprost 0.005% (Active Comparator): Latanoprost Ophthalmic Solution, 0.005% dosed once daily to both eyes (initial phase of trial)
  Interventions: Drug: Latanoprost 0.005% (initial phase of trial)
- NCX 470 0.1% (remainder of trial) (Experimental): NCX 470 Ophthalmic Solution, 0.1% dosed once daily to both eyes (chosen dose of NCX 470 to continue in remainder of trial)
  Interventions: Drug: NCX 470 0.1% (remainder of trial)
- Latanoprost 0.005% (remainder of trial) (Active Comparator): Latanoprost Ophthalmic Solution, 0.005% dosed once daily to both eyes (active comparator for remainder of trial)
  Interventions: Drug: Latanoprost 0.005% (remainder of trial)

INTERVENTIONS:
Drug: NCX 470 0.065% (initial phase of trial) — NCX 470 Ophthalmic Solution, 0.065% (initial phase of trial)
  Arms: NCX 470 0.065%
Drug: Latanoprost 0.005% (initial phase of trial) — Latanoprost Ophthalmic Solution, 0.005%
  Other Names: Latanoprost
  Arms: Latanoprost 0.005%
Drug: NCX 470 0.1% (initial phase of trial) — NCX 470 Ophthalmic Solution, 0.1%
  Arms: NCX 470 0.1%
Drug: NCX 470 0.1% (remainder of trial) — NCX 470 Ophthalmic Solution, 0.1%
  Arms: NCX 470 0.1% (remainder of trial)
Drug: Latanoprost 0.005% (remainder of trial) — Latanoprost Ophthalmic Solution, 0.005%
  Arms: Latanoprost 0.005% (remainder of trial)

SUMMARY:
The objective of this clinical study is to evaluate the safety and efficacy of NCX 470 Ophthalmic Solution in lowering intraocular pressure (IOP) in patients with ocular hypertension or open-angle glaucoma. In the adaptive dose selection phase of the trial, subjects will be randomized in a 1:1:1 ratio to one of two doses of NCX 470 (0.065% or 0.1%) or to latanoprost 0.005%. Following the selection of one dose of NCX 470, subjects will be randomized in a 1:1 ratio to the chosen dose of NCX 470 or to latanoprost 0.005%.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension in both eyes
* Qualifying IOP at 3 time points through the day at 2 visits following washout of IOP-lowering medication, if applicable
* Qualifying best-corrected visual acuity in each eye
* Ability to provide informed consent and follow study instructions

Exclusion Criteria:

* Narrow anterior chamber angles or disqualifying corneal thickness in either eye
* Clinically significant ocular disease in either eye
* Previous complicated surgery or certain types of glaucoma surgery in either eye
* Incisional ocular surgery or severe trauma in either eye within the past 6 months
* Uncontrolled systemic disease

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 691 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicox Ophthalmics, Inc., Study Director — Nicox Ophthalmics, Inc.
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 56 ophthalmologists' clinics in the US and 1 clinic in China. The first participant for the study was screened in June 2020 and the last participant exited the trial in September 2022.
Pre-assignment Details: Participants were consented and screened for eligibility. Subjects underwent a medication wash-out. Eligible subjects meeting IOP criteria were randomized to 1 of 3 groups. All participants dosed once daily in both eyes. After 30 subjects in all 3 arms completed 2 weeks on drug, a planned, Adaptive Analysis was performed. Based upon the results of this analysis, enrollment continued in the NCX 470 0.1% and latanoprost 0.005% groups and the NCX 0.065% arm was discontinued.
Groups:
- NCX 470 0.065%: NCX 470 Ophthalmic Solution, 0.065% dosed once daily to both eyes
- NCX 470 0.1%: NCX 470 Ophthalmic Solution, 0.1% dosed once daily to both eyes
- Latanoprost 0.005%: Latanoprost Ophthalmic Solution, 0.005% dosed once daily to both eyes
Period: Overall Study
Arm/Group | NCX 470 0.065% | NCX 470 0.1% | Latanoprost 0.005%
Started | 30 | 328 | 333
Completed | 27 | 314 | 316
Not Completed | 3 | 14 | 17
Not completed — Due to adaptive design | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 4
Not completed — Sponsor or IRB Decision | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 3
Not completed — Adverse Event | 0 | 8 | 6
Not completed — Other Reason | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A study eye was assigned based upon the baseline IOP collected at the Eligibility Visits. The primary efficacy analysis was performed on the study eye and the fellow was followed for safety.
Groups:
- Total: Total of all reporting groups
Arm/Group | NCX 470 0.065% | NCX 470 0.1% | Latanoprost 0.005% | Total
Number analyzed (Participants) | 30 | 328 | 333 | 691
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 168 | 174 | 353
  >=65 years | 19 | 160 | 159 | 338
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 200 | 188 | 405
  Male | 13 | 128 | 145 | 286
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 59 | 67 | 133
  Not Hispanic or Latino | 23 | 267 | 265 | 555
  Unknown or Not Reported | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 0 | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 9 | 110 | 109 | 228
  White | 20 | 212 | 216 | 448
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 328 | 332 | 690
  China | 0 | 0 | 1 | 1
Time-Matched IOP [Mean (Standard Deviation); unit: mmHg] — Baseline time-matched IOP is the average of the IOP at Eligibility 1 and Eligibility 2 Visits (study eye)
  mmHg
    Time-Matched IOP 8AM | 28.07 (2.286) | 28.28 (2.000) | 28.22 (2.011) | 28.19 (2.099)
    Time-Matched IOP 4PM | 25.15 (2.589) | 25.52 (2.455) | 25.40 (2.422) | 25.36 (2.489)

OUTCOME MEASURES:

1. Primary Outcome: Mean IOP Reduction From Time-Matched Baseline at the 8AM and 4PM Time-Points at Week 2, Week 6, and Month 3
Description: The analysis performed as part of the Adaptive Dose Phase of the study was to evaluate the efficacy and safety of both concentrations of NCX 470 compared to Latanoprost. The primary endpoint for the interim analysis was mean diurnal IOP. Subsequent to the interim analysis at Week 2, the NCX 470 0.065% arm was discontinued and the primary analysis only included NCX 470 0.1% vs Latanoprost. The primary efficacy outcome results are reported for the NCX 470 0.1% and Latanoprost 0.005% treatment groups at Week 2, Week 6, and Month 3. As prespecified in the Statistical Analysis Plan, mean change from baseline in time-matched IOP was not calculated for the 0.065% group.
  The study eye was defined as the eye with the highest mean diurnal intraocular pressure (IOP) value at baseline (or right eye if both eyes had the same IOP value at baseline). The fellow eye was followed for safety.
Time Frame: Baseline, Week 2, Week 6, and Month 3
Population: Participants used medication in both eyes for 3 months with 1 eye designated as study eye at baseline. The study eye was defined as the eye with the highest mean diurnal intraocular pressure (IOP) value at baseline (or right eye if both eyes had the same IOP value at baseline).
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | NCX 470 0.1% | Latanoprost 0.005%
Number analyzed (Participants) | 328 | 333
Number analyzed (eyes) | 328 | 333
mmHg
  Mean change from baseline - Week 2 8AM | -9.43 (3.443) | -8.85 (3.349)
  Mean change from baseline - Week 2 4PM | -8.01 (3.379) | -7.11 (3.330)
  Mean change from baseline - Week 6 8AM | -9.69 (3.129) | -9.33 (3.395)
  Mean change from baseline - Week 6 4PM | -8.18 (3.093) | -7.14 (3.283)
  Mean change from baseline - Month 3 8AM | -9.61 (3.196) | -9.39 (3.345)
  Mean change from baseline - Month 3 4PM | -8.00 (3.026) | -7.31 (3.296)
Statistical Analysis 1: Comparison: NCX 470 0.1% vs Latanoprost 0.005%; Test type: Non-Inferiority — Non-inferiority was concluded if the lower limit of the 95.1% CIs around the difference (NCX 470 minus latanoprost 0.005%) in mean IOP reduction from time-matched baseline in the study eye was greater than or equal to -1.5 mmHg at all time points and was greater than or equal to -1.0 mmHg at a majority of the time points; The primary efficacy assessment was the non-inferiority analysis of the difference in the treatment effect between NCX 470 and latanoprost 0.005% for mean IOP reduction from time-matched baseline at the 8AM and 4PM time-points; Mean Difference (Net) = 1.0, Standard Deviation 3.25 — The analysis assumed a true difference of 1.0 mmHg at the Week 2 time points and 1.25 mmHg at the Week 6 and Month 3 time points; a common standard deviation (SD) at each time-point of 3.25 mmHg; and a two-sided significance level of 4.9%

2. Secondary Outcome: Reduction From Baseline in Mean Diurnal IOP at Week 2, Week 6, and Month 3 in the Study Eye
Description: Subjects in the NCX 470 0.065% treatment group were discontinued at Week 2 based upon the results of the planned, interim analysis.
  Subjects in the NCX 470 0.1% and Latanoprost 0.005% treatment groups continued for 3 months.
  Participants used medication in both eyes for 3 months with 1 eye designated as study eye at baseline. The study eye was defined as the eye with the highest mean diurnal intraocular pressure (IOP) value at baseline (or right eye if both eyes had the same IOP value at baseline).
Time Frame: Baseline, Week 2, Week 6, and Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | NCX 470 0.1% | Latanoprost 0.005%
Number analyzed (Participants) | 328 | 333
Number analyzed (eyes) | 328 | 333
mmHg
  Change from Baseline to Week 2 in Mean Diurnal IOP | -8.82 (3.057) | -8.05 (3.020)
  Change from Baseline to Week 6 in Mean Diurnal IOP | -9.01 (2.758) | -8.34 (3.030)
  Change from Baseline to Month 3 in Mean Diurnal IOP | -8.90 (2.697) | -8.41 (2.952)

3. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAE) by Treatment Group in the Safety Population
Description: Safety and tolerability based on number subjects with treatment emergent ocular adverse events.
Time Frame: 3 months
Population: Safety population - all subjects who were randomized to treatment and received 1 dose of study medication.
Measure: Number; unit: numbers subjects with TEAEs
Arm/Group | NCX 470 0.065% | NCX 470 0.1% | Latanoprost 0.005%
Number analyzed (Participants) | 30 | 328 | 333
numbers subjects with TEAEs
  Any Ocular TEAEs | 13 | 113 | 58
  Any Non-Ocular TEAEs | 1 | 37 | 32
  Any serious Ocular TEAEs | 0 | 0 | 0
  Any serious Non-Ocular TEAEs | 0 | 4 | 3
  Any serious Ocular TEAEs related to study drug | 0 | 0 | 0
  Any serious Non-Ocular TEAEs related to study drug | 0 | 0 | 0

4. Secondary Outcome: Rate of Discontinuation
Description: Number of subjects discontinued from the study.
Time Frame: 3 months
Population: Subjects who were randomized to study drug and did not complete the study.
Measure: Count of Participants; unit: Participants
Arm/Group | NCX 470 0.065% | NCX 470 0.1% | Latanoprost 0.005%
Number analyzed (Participants) | 30 | 328 | 333
Participants | 3 | 14 | 17

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 90 days of dosing of study drug.
Arm/Group | NCX 470 0.065% | NCX 470 0.1% | Latanoprost 0.005%
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/328 | 2/333
Serious Adverse Events (participants affected / at risk) | 0/30 | 4/328 | 3/333
Other Adverse Events (participants affected / at risk) | 12/30 | 112/328 | 32/333
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NCX 470 0.065% (N=30) | NCX 470 0.1% (N=328) | Latanoprost 0.005% (N=333)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Systemic event
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Systemic event
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Systemic event
Corona Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) — Systemic event
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Systemic event
Transient ischemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Systemic event
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NCX 470 0.065% (N=30) | NCX 470 0.1% (N=328) | Latanoprost 0.005% (N=333)
Conjunctival hyperemia (Eye disorders) | 5 (5) | 36 (36) | 7 (7) — Ocular event
Ocular hyperemia (Eye disorders) | 1 (1) | 39 (39) | 11 (11) — Ocular event
Eye pruritus (Eye disorders) | 1 (1) | 17 (17) | 6 (6) — Ocular event
Instillation site pain (General disorders) | 5 (5) | 20 (20) | 8 (8) — Ocular event

LIMITATIONS AND CAVEATS:
This was a robust, international trial demonstrating the safety and efficacy of NCX 470 0.1% Ophthalmic Solution. A 2nd Phase 3 trial is on-going and the sponsor expects the results of the 2nd trial to be consistent with the results of this study. While this study was only 3 months in length, the 2nd trial is a 12-month study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT04445519/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT04445519/SAP_001.pdf